CLINICAL TRIAL: NCT00116168
Title: A Phase I, Open Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single-Dose Subcutaneous Administration of MEDI-528, a Humanized Monoclonal Anti-Interleukin-9 Antibody, in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single-Dose Subcutaneous Administration of MEDI-528
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP109
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — enokizumab

ARMS (4):
- MEDI-528 0.3 mg/kg (Experimental): MEDI-528 (0.3 mg/kg) administered as a single, subcutaneous (SC) dose
  Interventions: Biological: MEDI-528 0.3 mg/kg
- MEDI-528 1 mg/kg (Experimental): MEDI-528 (1 mg/kg) administered as a single, SC dose
  Interventions: Biological: MEDI-528 1 mg/kg
- MEDI-528 3 mg/kg (Experimental): MEDI-528 (3 mg/kg) administered as a single, SC dose
  Interventions: Biological: MEDI-528 3 mg/kg
- MEDI-528 9 mg/kg (Experimental): MEDI-528 (9 mg/kg) administered as a single, SC dose
  Interventions: Biological: MEDI-528 9 mg/kg

INTERVENTIONS:
Biological: MEDI-528 0.3 mg/kg — MEDI-528 (0.3 mg/kg) administered as a single, subcutaneous (SC) dose
  Arms: MEDI-528 0.3 mg/kg
Biological: MEDI-528 1 mg/kg — MEDI-528 (1 mg/kg) administered as a single, SC dose
  Arms: MEDI-528 1 mg/kg
Biological: MEDI-528 3 mg/kg — MEDI-528 (3 mg/kg) administered as a single, SC dose
  Arms: MEDI-528 3 mg/kg
Biological: MEDI-528 9 mg/kg — MEDI-528 (9 mg/kg) administered as a single, SC dose
  Arms: MEDI-528 9 mg/kg

SUMMARY:
A Phase I studyto evaluate the safety and tolerability of escalating subcutaneous (SC) doses of MEDI-528 in to healthy adult volunteers.

DETAILED DESCRIPTION:
The primary objective of this Phase I study is to evaluate the safety and tolerability of escalating single SC doses of MEDI-528 administered to healthy adult volunteers in four dose groups.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 19 up to, and including, 49 years of age at the time of the first dose of study drug
* Weight less than 89 kg
* Written informed consent obtained from the volunteer
* Healthy by medical history and physical examination
* Sexually active females, unless surgically sterile or at least two years post-menopausal or an FSH≥40 mIu/mL, must use an effective method of avoiding pregnancy (including oral, injectable, transdermal, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 3 months before the first dose of study drug, and must agree to continue using such precautions through the study period of 84 days. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active males, unless surgically sterile, must likewise use an effective method of birth control (condom or abstinence) and must agree to continue using such precautions through Study Day 84 after their dose of study drug.
* Use of common over-the-counter medications such as topical corticosteroids, decongestants, antihistamines, analgesics, and antacids is permitted unless, in the opinion of the investigator, it would interfere with either the volunteer's ability to complete the study or interpretation of the study results.
* Ability to complete the follow-up period of 84 days
* Willing to forego other forms of experimental treatment during the study period of 84 days
* Willing to forego vigorous activity 1 - 2 days before dosing, and before each study visit.

Exclusion Criteria:

* Acute illnesses or evidence of significant active infection, such as fever greater than or equal to 38.0 C (100.5°F) at the start of the study
* Use of prescription medications, other than oral contraceptives, in the 28-day period before Study Day 0
* Any blood donation or significant loss of blood within 6 months of time of entry into the study
* History of immunodeficiency or receipt of immunosuppressive drugs
* History of allergy or reaction to any component of the MEDI-528 formulation
* History of substance abuse that, in the opinion of the investigator, may compromise the ability of the study subject to complete the study and follow-up period
* Evidence of any systemic disease, neurologic abnormality, lymphadenopathy, or splenomegaly upon physical examination
* Evidence of infection with hepatitis A, B, or C virus or HIV-1
* Receipt of immunoglobulins or blood products within 60 days of entering the study
* Receipt of any investigational drug therapy or standard vaccine therapy, other than vaccination for influenza, within 60 days of the first dose of study drug through Study Day 84 (use of licensed agents for indications not listed in the package insert is permitted)
* Receipt of MEDI-528 in any previous clinical study
* At Screening (must be within 21 days before study dose administration) any of the following: Hgb, total WBC, platelet count, Na, K, C1, CO2, AST, ALT, BUN, glucose, amylase, lipase, creatinine, or troponin out of the normal range; other abnormal laboratory values in the screening panel that, in the opinion of the principal investigator, are judged to be clinically significant
* Clinically significant abnormality, as determined by the investigator, on 12-lead electrocardiogram at the time of initial screening
* Clinically significant abnormalities noted on baseline brain MRI
* Elective surgery planned during the study period through Study Day 84
* Pregnancy (sexually active females must have a negative serum pregnancy test on the day of the first dose of study drug, before dosing)
* Nursing mother
* The presence of any condition or concern which, in the opinion of the investigator, may interfere with the conduct or interpretation of the study.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara White, M.D., Study Director — MedImmune LLC
Locations (2):
- United States (2):
  - MDS Pharma Services, New Orleans, Louisiana
  - MDS Pharma Services, Lincoln, Nebraska

REFERENCES:
- [Derived] White B, Leon F, White W, Robbie G. Two first-in-human, open-label, phase I dose-escalation safety trials of MEDI-528, a monoclonal antibody against interleukin-9, in healthy adult volunteers. Clin Ther. 2009 Apr;31(4):728-40. doi: 10.1016/j.clinthera.2009.04.019. PMID 19446146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 29 participants provided written informed consent and participated in the study at 2 sites in the United States of America between 10Jun2005 and 18Apr2006.
Pre-assignment Details: Eligible participants received MEDI-528 in an open-label manner.
Period: Overall Study
Arm/Group | MEDI-528 0.3 mg | MEDI-528 1 mg | MEDI-528 3 mg | MEDI-528 9 mg
Started | 6 | 11 | 6 | 6
Completed | 0 | 6 | 6 | 6
Not Completed | 6 | 5 | 0 | 0
Not completed — Lost to Follow-up | 6 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI-528 0.3 mg | MEDI-528 1 mg | MEDI-528 3 mg | MEDI-528 9 mg | Total
Number analyzed (Participants) | 6 | 11 | 6 | 6 | 29
Age Continuous [Mean (Standard Deviation); unit: Years] | 27.2 (8.7) | 25.2 (9.7) | 34.7 (7.8) | 33.2 (13.9) | 29.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 3 | 14
  Male | 2 | 7 | 3 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Number of participants experiencing adverse events (includes both adverse events and serious adverse events)
Time Frame: Days 0 - 84
Population: All subjects who received MEDI-528 (no safety information was available for 5 subjects in the 1.0 mg/kg group due to Hurricane Katrina)
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 5 | 4 | 6 | 6

2. Primary Outcome: Incidence of Abnormal Troponin Levels
Description: Number of participants with troponin levels greater than upper limit of normal
Time Frame: Days 0, 1, 7, 14, and 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Clinically Significant Changes From Baseline in Neurologic Exam
Description: Number of participants with clinically significant changes from baseline in neurologic exam
Time Frame: Days 0, 7, 14, 21, 28, 42, and 84
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Changes From Baseline in the Day 28 Magnetic Resonance Imaging (MRI) of the Brain
Description: Number of participants with changes from baseline in the Day 28 MRI of the brain
Time Frame: Days 0 and 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 1 | 1 | 1

5. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of participants experiencing serious adverse events
Time Frame: Days 0 - 84
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) to MEDI-528
Description: Number of participants with ADA to MEDI-528
Time Frame: Days 0, 14, 28, 42, and 84
Population: All subjects who received MEDI-528 (no safety or ADA information was available for 5 subjects in the 1.0 mg/kg group due to Hurricane Katrina). Partial ADA information was available in the 0.3 mg/kg group (Day 0 and 14, n=5; Day 28, n=2; Day 42 and 84, n = 0)
Measure: Number; unit: Participants
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 5 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Time to Observed Maximum Serum Concentration (Tmax)
Description: Tmax of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: All subjects who received MEDI-528 (no safety information was available for 5 subjects in the 1.0 mg/kg group due to Hurricane Katrina). Two subjects in the 0.3 mg/kg group had no blood samples for pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 4 | 6 | 6 | 6
Days | 5.51 (1.90) | 4.17 (1.60) | 4.50 (1.52) | 5.00 (1.90)

8. Secondary Outcome: Observed Maximum Serum Concentration (Cmax)
Description: Cmax of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 4 | 6 | 6 | 6
Micrograms per milliliter | 2.83 (0.73) | 14.48 (6.68) | 23.00 (5.62) | 82.50 (19.64)

9. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Last Measurable Concentration [AUC(0-t)]
Description: AUC(0-t) of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Micrograms times day per milliliter
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 4 | 6 | 6 | 6
Micrograms times day per milliliter | 18.47 (10.26) | 329.7 (113.72) | 923.27 (226.71) | 3053.34 (908.30)

10. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Infinity [AUC(0-infinity)] of MEDI-528
Description: AUC(0-infinity) of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Microgram times day per milliliter
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 6
Microgram times day per milliliter | 40.78 (0.34) | 667.68 (201.99) | 1287.31 (413.92) | 3770.06 (1396.66)

11. Secondary Outcome: Percent of Total Area Under the Concentration Curve Extrapolated From Last Measurable Time to Infinity [AUC(Ext)]
Description: AUC(ext) of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 6
Percent | 33.32 (6.26) | 50.90 (13.82) | 26.05 (9.16) | 16.61 (8.97)

12. Secondary Outcome: Total Body Clearance (CL)
Description: CL of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liter per day
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 6
Liter per day | 0.49 (0.00) | 0.12 (0.05) | 0.19 (0.10) | 0.20 (0.09)

13. Secondary Outcome: Half-life (T1/2)
Description: T1/2 of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 6
Days | 6.47 (0.85) | 86.85 (19.86) | 44.43 (11.48) | 33.44 (11.32)

14. Secondary Outcome: Apparent Extravascular Terminal Phase Volume of Distribution (Vz/F)
Description: Vz/F of MEDI-528
Time Frame: Days 0, 1, 2, 3, 4, 5, 7, 10, 14, 21, 28, 42, and 84
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | MEDI-528 0.3 mg/kg | MEDI-528 1 mg/kg | MEDI-528 3 mg/kg | MEDI-528 9 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 6
Liters | 4.58 (0.64) | 14.57 (8.61) | 10.91 (1.21) | 8.65 (1.40)

ADVERSE EVENTS:
Time Frame: Days 0-84
Description: No safety information was available for 5 subjects in the 1.0 mg/kg group due to Hurricane Katrina.
Arm/Group | MEDI-528 0.3 mg | MEDI-528 1 mg | MEDI-528 3 mg | MEDI-528 9 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-528 0.3 mg (N=6) | MEDI-528 1 mg (N=6) | MEDI-528 3 mg (N=6) | MEDI-528 9 mg (N=6)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood chloride increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Protein urine present (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.